CLINICAL TRIAL: NCT07074743
Title: Evaluate the Feasibility and Effectiveness of a Community-based Care Bundle in Managing and Preventing Pressure Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other); Singapore Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022/2406_CAPIcarebundle
Record Dates: First submitted 2025-06-29; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Pressure Injuries; Caregiver; Community Dwelling Older Adult
Keywords: pressure injuries; community nursing; care bundle
MeSH Terms: conditions — Pressure Ulcer | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait-list (Active Comparator): The wait-list group will receive routine care during the first six weeks and at seven weeks, the index PI will be restaged and if patient is still having PI- the PI care bundle will be provided for the next six weeks. However, PI care bundle can also be initiated if the index PI advances to higher stage had increased pain over PI site or when there is deterioration of the index PI at any point during the weekly follow up.
  Providing PI care bundle to wait-list control group after 6 week ensures ethical care while maintaining study integrity.
  Interventions: Other: Wait-list
- Community-based PI care bundle (Experimental): The community-based PI care bundle follows the aSSKINg model and is delivered in addition to routine care for six weeks.
  Interventions: Other: community-based PI care bundle

INTERVENTIONS:
Other: community-based PI care bundle — The PI care bundle follows the aSSKINg model and is delivered in addition to routine care. Key components include:
  Assessment Pre-discharge evaluation Ongoing skin, nutrition, and hydration monitoring Caregiver training for home assessment Equipment and Resources
  Customized provision of necessary devices based on needs:
  Sliding sheets Repositioning cushions Skin barriers Moisturizers Pressure-relieving overlays Alternating air mattresses Implementation Caregivers demonstrate device usage competency Documentation checklist for monitoring Regular follow-up by community nurses Professional Support Community nurses trained by PI specialists Standardized care protocols Regular effectiveness assessment
  All participants receive routine care including:
  Pre-discharge nutrition assessment Dietician referral if needed Educational materials Basic wound care referrals Hospital-to-home team support for complex cases The intervention provides structured, comprehensive support beyond standard care.
  Arms: Community-based PI care bundle
Other: Wait-list — During hospitalisation:
  Patient's nutritional status assessed. Referred to a dietician before discharge if needed. Nurse assesses caregiver training needs and arranges training if required.
  At discharge:
  Patients receive PI educational pamphlets (hardcopy or softcopy). Emphasis on regular repositioning, skin inspection, proper nutrition, and hydration.
  Patients with PI wounds:
  Referred to home nursing or polyclinics for wound care. Only those with complex PI (stage >3) receive up to two follow-ups by the H2H care team.
  H2H team supports general care transition, not PI-specific follow-up alone. Any signs of PI deterioration will be monitored weekly throughout the waiting period for safety and ethical considerations.
  If the index PI advances to a higher stage and reports increased pain after a week, the investigator will refer them to a community wound care nurse and record this as a deterioration and will start PI care bundle
  Other Names: routine care; usual care
  Arms: Wait-list

SUMMARY:
Community-acquired pressure injuries are pressure injuries that developed outside of hospital, typically in the patient's own home environment. Pressure injuries (PI) used to be commonly known as bedsores or pressure ulcers.

The goal of this clinical trial is to evaluate if a community-based pressure injury (PI) care bundle is effective in treating and preventing pressure injuries in home settings. It will also assess how feasible it is to implement this care bundle in Singapore's community care context.

The main questions it aims to answer are:

1. Does the PI care bundle help improve pressure injury healing (shown by at least a 3-point reduction on the PUSH score)?
2. Can the care bundle prevent the development of new pressure injuries?
3. How well do caregivers learn and apply PI care knowledge after receiving the educational intervention?
4. How practical and acceptable is this care bundle for use in home settings?

The investigators will compare the PI care bundle to routine care (control group) to see if the care bundle works better for managing pressure injuries at home. Success will be measured using the PUSH tool, which scores pressure injuries from 0 (completely healed) to 17 (most severe). A reduction of at least 3 points on this scale will indicate meaningful improvement.

Participants and their caregivers will:

Be split into two groups - one group will use the new care plan (receive the PI care bundle), and the other will continue with their routine care.

Have their pressure injuries checked regularly for 6 weeks. Have their caregivers learn about pressure injury care. Answer questions about how well the care plan works for them.

The investigator hopes this study will help find better ways to treat or prevent pressure injuries at home and support the caregivers at home.

DETAILED DESCRIPTION:
STUDY DESIGN and METHODOLOGY

This is a randomized controlled trial evaluating a community-based pressure injury (PI) care bundle versus routine care. The study employs a waitlist-control design with a 6-week intervention period.

OUTCOME MEASUREMENTS

Primary Outcome:

* Clinical improvement measured using the Pressure Ulcer Scale for Healing (PUSH) tool.
* Minimum clinically meaningful effect size established as 3-point reduction on PUSH score.
* PUSH scoring ranges from 0 (healed) to 17 (most severe)

Secondary Outcomes:

* Incidence of new pressure injuries
* Caregiver Knowledge, Attitudes, and Practices (KAP) assessment

Feasibility metrics including:

* Implementation appropriateness
* Intervention acceptability
* Protocol fidelity
* Participation and retention rates
* Adherence to prescribed prevention measures

TECHNICAL COMPONENTS OF CARE BUNDLE

The intervention group will receive:

* Using the aSSKINg framework, the investigators have co-design the content of PI prevention and management with the community nurses, WOC nurses and caregivers.
* Delivered a structured caregiver education program- tailored to the patient and caregiver needs.
* Weekly check in by the study team or community nurses
* Documentation and tracking tools using electronic wound imaging system.

DATA COLLECTION AND ANALYSIS

Standardized assessment tools for PI staging- PI staging follows National Pressure Injury Advisory Panel (NPIAP) standardized system.

Validated KAP questionnaires Feasibility assessment metrics Protocol adherence monitoring Dropout rate tracking

Statistical analysis comparing intervention versus control outcomes.

The study design incorporates rigorous methodology to evaluate both clinical effectiveness and implementation feasibility in the community setting, with specific attention to the unique challenges of home-based PI care management.

ELIGIBILITY:
Inclusion Criteria

* adult patients discharged from SGH with existing PI (any stages according to NPIAP and on any part of the body)
* have a family caregiver or FDH who will be managing the PI upon discharge
* patients will be discharged to home
* living within the SGH nursing community zones

Exclusion Criteria

* previous or existing participation in this trial
* palliative or dying patients
* planned discharge to a nursing home or other hospital
* mobile inpatient care@home service
* patient or next-of-kin who refused to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pressure injury healing | at 6 weeks post randomisation
  The proportion of community-dwelling adults who achieve a reduction of at least 3 points on the PUSH score of the index PI at six weeks. The PUSH tool, with a range from 0 (healed) to 17 (worst score), provides a continuous outcome measure. The investigators have set a 3-point reduction as the minimum clinically meaningful effect size for this study.

SECONDARY OUTCOMES:
Caregiver's Knowledge, Attitude and Practice (KAP) | 6 weeks post randomisation
  Changes in caregivers' KAP scores will be compared at baseline and six-week scores between groups.
  Knowlege domain: 12 MCQs, lowest score 0 to highest 12. A cut of point of 65% will be considered sufficient.
  Attitude domain: consist of 9 statements on PI prevention, participants will be asked to indicate the extent of their agreement from strongly agree (score 4) and strongly disagree (score 1). The sum score range 9 to 36; a higher score indicate more positive attitude.
  Practice domain: consist of 12 statements PI preventive care measures. Using a Likert scale: never to always. The sum of score range 12 to 48. A higher score indicate better PI practice.

OTHER OUTCOMES:
Feasibility of the community-based PI care bundle | At completion of the study, i.e. at the end of 6 weeks.
  Feasibility will be assessed using acceptability indicator:
  (1) Acceptability, measured by patient and caregiver satisfaction using a self-validated questionnaire, with success defined as high satisfaction (>70%), high participation (>70%), and low dropout rates (<20%);
Feasibility of the community-based PI care bundle | At completion of the study, i.e. at the end of 6 weeks.
  Feasibility will be assessed using adherence indicator:
  (2) Adherence, measured as the proportion of patients and caregivers following recommended PI prevention measures, with a target of ≥70%
Feasibility of the community-based PI care bundle | At completion of the study, i.e. at the end of 6 weeks.
  Feasibility will be assessed using fidelity indicator:
  (3) Fidelity, evaluated through audits of care bundle implementation, with success defined as achieving ≥80%.

CONTACTS AND LOCATIONS:
Overall Officials: Fazila Aloweni, MSci, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: ICF
Time Frame: Beginning 1 months and ending 1 years after the publication of results
Access Criteria: The PI's research office will review the request